CLINICAL TRIAL: NCT01700023
Title: Pilot-study HI-SENS: Innovative Sensor Technology to Quantify Cardiac Control Mechanisms in Heart Failure
Brief Title: 3-dimensional Sensor Technology to Quantify Leg-edema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Collaborators: AIT Austrian Institute of Technology GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: 24-536 ex 11/12
Record Dates: First submitted 2012-09-30; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: ADHF
Keywords: acute heart failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with leg-edema: patients with decompensated heart failure presenting with leg-edema

SUMMARY:
The purpose of the study is two-fold:

1. to test 3-dimensional reconstruction of leg-edema in patients hospitalized for acute heart failure with leg-edema.
2. to measure changes in QRS-morphology in a simulation of conventional blood-pressure measurement in patients hospitalized for acute heart failure.

DETAILED DESCRIPTION:
Leg-edema are common in patients with worsening heart failure. Apart from using a measuring tape there is no standardized tool to quantify leg-edema. Consequently, in patents with heart failure early detection of leg-edema is quite difficult.

From earlier pacemaker-studies it has been shown that an increase of afterload changes ECG-signals. Currently it is unknown how simple diagnostic procedures such as measuring blood-pressure affect QRS-morphology in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* hospitalization for worsening heart failure
* age greater than 18 years
* ability to stand without help from others
* informed consent

Exclusion Criteria:

* leg-edema of non-cardiac origin (venous, lymphatic)
* dialysis shunt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized for decompensated heart failure with leg-edema
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2012-09; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
accuracy of 3-dimensional measurements | 10 days
  the 3-D camera will record changes in leg-shape around the ankles that result from reabsorption of fluid. These changes will be compared with changes in leg-circumference using a measuring tape

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich M Fruhwald, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University, Graz, Austria